CLINICAL TRIAL: NCT00004753
Title: Long-Term Study of Cerebral Glucose Metabolism in Huntington's Disease
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of California, Los Angeles (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11677; UCLA-90063784
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Huntington's Disease
Keywords: Huntington's disease; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Huntington Disease; Neurologic Manifestations; Mental Disorders; Rare Diseases

SUMMARY:
OBJECTIVES: I. Correlate clinical outcome with cerebral glucose metabolism in patients with Huntington's disease (HD) and their at-risk relatives.

II. Evaluate the efficacy of cerebral glucose metabolism in observing the pathophysiologic development of HD, monitoring responses to experimental therapy, and predicting HD genotype.

III. Identify, define, and describe the natural history of pathophysiologic lesions in HD.

IV. Characterize the genotypic and phenotypic expression of the HD gene.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Participants are screened for Huntington's disease, including cerebral glucose metabolism assessment and genetic testing.

Studies include a detailed family history and neurologic, psychometric, and neurobehavioral evaluations. Imaging includes positron emission tomography with fluorodeoxyglucose and brain magnetic resonance imaging.

A genotype assessment is performed; genetic results are not disclosed to patients or relatives.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Documented family history of Huntington's disease (HD)
* Symptomatic HD: chorea required
* At-risk for HD: no detectable systemic or oculomotor abnormality
* Age-matched control subjects
* No history of inherited neurological disease
* No general or neurologic abnormality

--Prior/Concurrent Therapy--

At least 4 weeks since other HD treatment, e.g.:

* Haloperidol
* Benzodiazepine
* Other tranquilizers or neuroleptics

--Patient Characteristics--

* No pregnant women

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 1993-08

CONTACTS AND LOCATIONS:
Overall Officials: John C. Mazziotta, Study Chair — University of California, Los Angeles